CLINICAL TRIAL: NCT00005356
Title: Novel Hemostatic Cardiac Risk Factors in Framingham
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4242; R01HL048157 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Death, Sudden, Cardiac; Myocardial Infarction; Thrombosis; Atherosclerosis; Carotid Artery Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Death, Sudden, Cardiac; Myocardial Infarction; Thrombosis; Atherosclerosis; Carotid Artery Diseases

SUMMARY:
To investigate hemostatic variables in relation to cardiovascular risk in the Framingham Offspring Study cohort.

DETAILED DESCRIPTION:
BACKGROUND:

Elevation of platelet reactivity plasminogen activator inhibitor, fibrinogen, von Willebrand's factor, and factor VII have been reported to increase myocardial infarction risk. Myocardial infarction and sudden cardiac death are more frequent in the morning when platelet activity is increased and fibrinolysis is decreased. Reduction of recurrent myocardial infarction by aspirin and coumadin suggests causal roles for platelet activity and coagulation. Increases in viscosity and decreases in anti-thrombin III and Protein C have been linked with increased thrombosis. Despite these findings, a coherent picture of these disparate hemostatic indices as cardiac risk factors has yet to emerge.

DESIGN NARRATIVE:

Platelet reactivty, plasminogen activatator inhibitor, fibrinogen, von Willebrand's factor, factor VII, and other hemostatic risk factors were measured in all 4,000 subjects of the Framingham Offspring Study. The data were combined with the regularly collected Framingham data to: determine the relationships between hemostatic factors and carotid atherosclerosis as assessed by ultrasound; determine the relationship between hemostatic factors and the traditional cardiac risk factors; and determine if hemostatic risk factors independently predict myocardial infarction and cardiac death.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-07; Study Completion 1998-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Tofler — Beth Israel Deaconess Medical Center

REFERENCES:
- [Background] Welty FK, Mittleman MA, Wilson PW, Sutherland PA, Matheney TH, Lipinska I, Muller JE, Levy D, Tofler GH. Hypobetalipoproteinemia is associated with low levels of hemostatic risk factors in the Framingham offspring population. Circulation. 1997 Feb 18;95(4):825-30. doi: 10.1161/01.cir.95.4.825. PMID 9054738
- [Background] Rosito GB, Tofler GH. Hemostatic factors as triggers of cardiovascular events. Cardiol Clin. 1996 May;14(2):239-50. doi: 10.1016/s0733-8651(05)70277-0. PMID 8724556
- [Background] Poli KA, Tofler GH, Larson MG, Evans JC, Sutherland PA, Lipinska I, Mittleman MA, Muller JE, D'Agostino RB, Wilson PW, Levy D. Association of blood pressure with fibrinolytic potential in the Framingham offspring population. Circulation. 2000 Jan 25;101(3):264-9. doi: 10.1161/01.cir.101.3.264. PMID 10645922
- [Background] Meigs JB, Mittleman MA, Nathan DM, Tofler GH, Singer DE, Murphy-Sheehy PM, Lipinska I, D'Agostino RB, Wilson PW. Hyperinsulinemia, hyperglycemia, and impaired hemostasis: the Framingham Offspring Study. JAMA. 2000 Jan 12;283(2):221-8. doi: 10.1001/jama.283.2.221. PMID 10634338
- [Background] Gebara OC, Mittleman MA, Sutherland P, Lipinska I, Matheney T, Xu P, Welty FK, Wilson PW, Levy D, Muller JE, et al. Association between increased estrogen status and increased fibrinolytic potential in the Framingham Offspring Study. Circulation. 1995 Apr 1;91(7):1952-8. doi: 10.1161/01.cir.91.7.1952. PMID 7895352